CLINICAL TRIAL: NCT00870558
Title: Adjuvant Treatment by Intra-arterial Injection of Lipiodol-labeled Iodine-131 in Preventing Recurrence of Hepatocellular Carcinoma After Curative Treatment
Brief Title: Iodine I 131 Ethiodized Oil in Preventing Recurrent Cancer in Patients Who Have Undergone Treatment for Liver Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000626727; HCL-2004-348-3; INCA-RECF0436; HCL-LIPIODOL
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2009-04

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Ethiodized Oil

ARMS (2):
- Arm I (Experimental): Patients receive an intra-arterial infusion of iodine I 131 ethiodized oil.
  Interventions: Radiation: iodine I 131 ethiodized oil
- Arm II (Placebo Comparator): Patients receive an intra-arterial infusion of unlabeled ethiodized oil.
  Interventions: Drug: ethiodized oil

INTERVENTIONS:
Drug: ethiodized oil — Given as an intra-arterial infusion
  Arms: Arm II
Radiation: iodine I 131 ethiodized oil — Given as an intra-arterial infusion
  Arms: Arm I

SUMMARY:
RATIONALE: Iodine I 131 ethiodized oil may help prevent or delay the recurrence of cancer. It is not yet known whether iodine I 131 ethiodized oil is more effective than non-radiolabeled ethiodized oil in preventing recurrent cancer in patients who have undergone treatment for liver cancer.

PURPOSE: This randomized phase III trial is studying iodine I 131 ethiodized oil to see how well it works compared with non-radiolabeled ethiodized oil in preventing recurrent cancer in patients who have undergone treatment for liver cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether treatment with adjuvant intra-arterial iodine I 131 ethiodized oil reduces the percentage of tumor recurrence in patients with curatively treated hepatocellular carcinoma.

Secondary

* Evaluate the overall and recurrence-free survival of these patients.
* Evaluate the deterioration of liver function in these patients.
* Evaluate the toxicity of intra-arterial iodine I 131 ethiodized oil in these patients.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive an intra-arterial infusion of iodine I 131 ethiodized oil.
* Arm II: Patients receive an intra-arterial infusion of unlabeled ethiodized oil.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hepatocellular carcinoma (HCC)

  * Alpha-fetoprotein < 20 ng/mL
* Must have undergone curative treatment for HCC within the past 8-20 weeks, including 1 of the following:

  * Curative resection
  * Alcohol ablation, radiofrequency ablation, or cryotherapy (for 1 or 2 nodules < 5 cm in diameter)
* No ascites
* No other intrahepatic involvement or nodule progression as assessed by ultrasound
* No extrahepatic metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* ANC ≥ 1,500/mm³
* Platelet count ≥ 50,000/mm³
* Bilirubin ≤ 51 μmol/L
* Creatinine ≤ 120 μmol/L
* Not pregnant or nursing
* Negative pregnancy test
* Child-Pugh score < 8 (class B)
* No decompensated cirrhosis
* No encephalopathy
* No uncontrolled bleeding
* No portal thrombosis, right- or left-branch thrombosis, extrahepatic thrombosis, or portal reflux by doppler or CT scan
* No unstable medical or surgical disease
* No contraindication to vascular arteriography
* No history of complications after injection of iodine contrast agents
* Not incarcerated

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* No prior hormonal treatment, including tamoxifen and somatostatin analogs
* No prior systemic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-06; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Tumor recurrence at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Dumortier, MD — Hopital Edouard Herriot - Lyon
Locations (1):
- Hopital Edouard Herriot - Lyon, Lyon, France